CLINICAL TRIAL: NCT00283179
Title: Efficacy and Safety of Aripiprazole in the Treatment of Acutely Relapsed Patients With Schizophrenia or Schizoaffective Disorder With Risperidone as an Active Control
Brief Title: Aripiprazole in the Treatment of Acutely Relapsed Patients With Schizophrenia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Taiwan Otsuka Pharm. Co., Ltd (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 31-02-A01
Record Dates: First submitted 2006-01-26; First posted 2006-01-27 (Estimated); Last update posted 2008-05-15 (Estimated); Status verified 2006-01

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: Aripiprazole; Risperidone; Schizophrenia; Schizoaffective disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Aripiprazole; Risperidone

INTERVENTIONS:
Drug: Aripiprazole
Drug: Risperidone

SUMMARY:
To evaluate the efficacy, safety and tolerability of aripiprazole in the treatment of acutely relapsed patients with diagnoses of schizophrenia or schizoaffective disorder with risperidone as an active control.

DETAILED DESCRIPTION:
Medical treatment of schizophrenia uses antipsychotic drugs, which ameliorate the acute episodes and probably prevent or decrease the risk of occurrence of new episodes. Most antipsychotics share the ability to block postsynaptic dopaminergic receptors of the D2 subtype.

The typical antipsychotics (such as haloperidol and chlorpromazine) ameliorate acute episodes and possibly prevent or decrease the risk of occurrence of new episodes, but they have minimal effectiveness against negative symptoms, mood symptoms, and cognitive impairment, which often lead to poor social functioning. Its full Dopamine antagonism is often associated with a number of well-recognized debilitating side effects. One example is EPS. A new class of antipsychotics, the atypical agents (such as clozapine, risperidone, olanzapine), became available starting in the late-1980s. Their mode of action affects both the serotonin and dopamine (DA) receptors. They are better tolerated than the typical antipsychotics with regard to EPS, except at higher doses. The improvement in the side effect profile seen with the atypical antipsychotics is accompanied by efficacy against positive symptoms and perhaps some improvement in efficacy against negative symptoms. Although they offer better efficacy and lower rates of EPS compared to typical agents, they are associated with other side effects that may be of clinical concern. For example, olanzapine and clozapine have an increased incidence of weight gain and diabetes mellitus, risperidone is associated with hyperprolactinemia, and ziprasidone is associated with ECG QT interval prolongation. In addition to tolerability issues, a significant proportion of patients still do not adequately respond to these newer agents. A need still exists for efficacious alternatives that demonstrate improved tolerability and side effect profiles so as to enhance treatment compliance and long-term functioning.

Aripiprazole is a novel DA-serotonin stabilizer approved in U.S. for the management of schizophrenia. The unique mode of action of aripiprazole translates into efficacy against psychotic symptoms and a more favorable safety profile than current treatment. Its introduction will clearly provide patients and their families with a much-needed alternative to the antipsychotics currently available.

This study further examined the efficacy and safety of aripiprazole in patients having acute relapse of schizophrenia or schizoaffective disorder in Taiwan. The duration of this study was 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis: Schizophrenia or schizoaffective disorder, in an acute relapse.
* Duration of present episode/relapse: Randomization to this study occurred no more than four weeks following the day of initiation of any treatment for the last episode/relapse.
* Age: 18 to 65 years.
* Gender: Males and females (females of childbearing potential had a negative serum pregnancy test from screening visit, used acceptable contraception, and were not pregnant or lactating).
* Response to previous antipsychotic agents: Patients had responded to previous antipsychotic medication
* Current antipsychotic treatment: Prior to beginning the placebo-washout, patients had not been treated with a long-acting antipsychotic within the time required for one cycle of treatment with that long-acting antipsychotic, plus one week. Patients who had been treated with a long-acting antipsychotic within less than this time period might be enrolled in the study, providing they were judged by the investigator to be clearly clinically deteriorating.
* Positive and Negative Syndrome Scale scores: Patients had a total PANSS score of at least 60. In addition, patients had a score of at least 4 on any two of the four PANSS items that constitute a psychotic items subscale.
* Compliance with the protocol: Patients were rated reliably on the battery of psychiatric and movement rating scales required by the protocol.
* Informed Consent: Patients eligible to enter the study signed an informed consent form prior to the initiation of any study procedures.

Exclusion Criteria:

* Patients who, in the opinion of the investigator, had serious suicidal ideation or patients who were liable to serious suicide attempt, by clinical judgment.
* Patients presented with a first episode of schizophrenia or schizoaffective disorder
* Patients who had any of the following neurological diagnoses, whether under treatment or not, whether stable or not: migraine, epilepsy, Parkinson's disease, Alzheimer's disease, multiple sclerosis, residual of stroke, transient cerebral ischemic attacks, 'cerebral palsy' or any condition that required intermittent or maintenance treatment, or which was manifested by any abnormality on neurological examination.
* Patients who continued to take, or who potentially needed to take, during the double-blind portion of this study, any of the following concomitant medications, which could cause unwanted drug-to-drug interactions or which could confound the analysis of antipsychotic effectiveness of the randomly assigned study drug: carbamazepine, valproic acid or sodium valproate or divalproate sodium, lithium carbonate or lithium citrate.
* Patients who failed to withdraw from fluoxetine treatment at least 28 days prior to screening, if on treatment with fluoxetine.
* Patients with any gastrointestinal resection, stomach stapling, or any other condition that may impair the absorption of the study medication.
* Patients who had positive result in the urine screen for drugs of abuse (except for cannabis or medically-prescribed analgesics or benzodiazepines.)
* Patients who met the DSM-IV criteria for psychoactive substance dependence or patients with a history of substance or alcohol dependence within one month prior to the beginning of the study.
* Patients had any somatic condition whose symptoms or physical signs could be misinterpreted as signs or symptoms of schizophrenia or as adverse effects from antipsychotic medications.
* Patients with any acute or unstable medical condition.
* Patients who had taken an investigational drug within the four weeks, which preceded the start of placebo washout.
* Patients who were treatment-resistant.
* Patients who continued to take, or who potentially needed to take, during this study, any medication or substance that is known to be an inhibitor of the microsomal enzyme CYP2D6, or an inhibitor or a substrate of the microsomal enzyme CYP3A4.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2004-03; Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
PANSS-total score

SECONDARY OUTCOMES:
PANSS-positive score, PANSS-negative score, CGI-severity score, CGI-improvement score, and safety/tolerability.

CONTACTS AND LOCATIONS:
Overall Officials: Tzung-Jeng Hwang, M.D., M.P.H., Principal Investigator — National Taiwan University Hospital; Hung-Yu Chan, M.D., Principal Investigator — Taoyuan Psychiatric Center, Ministry of Health and Welfare, Executive Yuan, R.O.C. Taiwan; Wei-Wen Lin, M.D., Ph.D., Principal Investigator — Tri-Service General Hospital; Shih-Ku Lin, M.D., Principal Investigator — Taipei City Psychiatric Center; Tung-Ping T. Su, M.D., Principal Investigator — Taipei Veterans General Hospital, Taiwan; Hai-Gwo Hwu, M.D., Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Result] Chan HY, Lin WW, Lin SK, Hwang TJ, Su TP, Chiang SC, Hwu HG. Efficacy and safety of aripiprazole in the acute treatment of schizophrenia in Chinese patients with risperidone as an active control: a randomized trial. J Clin Psychiatry. 2007 Jan;68(1):29-36. doi: 10.4088/jcp.v68n0104. PMID 17284127